CLINICAL TRIAL: NCT03038854
Title: Effects of Milk Intake on Nutrient Status and Neurocognitive Development in Toddlers: a Partially Randomized and Controlled Trial
Brief Title: Growing Up Milk (GUM) Intake and Nutrient Status of Toddlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 14.16.INF
Record Dates: First submitted 2017-01-25; First posted 2017-02-01 (Estimated); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Healthy
MeSH Terms: interventions — Milk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test GUM (Experimental): This group will drink a test toddler growing up milk (GUM) with higher amounts of key nutrients
  Interventions: Other: Test GUM
- Standard GUM (Active Comparator): This group will drink a standard toddler growing up milk (GUM)
  Interventions: Other: Standard GUM
- Comparator Group (Placebo Comparator): This group will drink liquid full fat cows' milk
  Interventions: Other: Cows' milk
- Population Group (No Intervention): This group will eat and drink their usual foods with no interventions.

INTERVENTIONS:
Other: Test GUM — Growing up milks (GUMs) are milk-based drinks with vitamins and minerals for toddlers and pre-school children.
  Other Names: Growing up milk
  Arms: Test GUM
Other: Standard GUM — Growing up milks (GUMs) are milk-based drinks with vitamins and minerals for toddlers and pre-school children.
  Other Names: Growing up milk
  Arms: Standard GUM
Other: Cows' milk — Homogenized store-bought full fat cow's milk.
  Arms: Comparator Group

SUMMARY:
The purpose of this study is to determine the nutritional and cognitive effects of consuming Growing Up Milks (GUMs) and cow's milk.

DETAILED DESCRIPTION:
Single-site, double blind, partially randomized, controlled, 4-arm parallel group clinical trial. The purpose of this study is to determine if consuming nutrient enriched growing up milk improves the nutrition status and cognitive performance in healthy toddlers.

ELIGIBILITY:
Inclusion Criteria:

1. Having obtained his/her parent's(s') or his/her legal guardian written informed consent and signed and dated informed consent.
2. Age 17 - 18 months at enrolment.
3. Singleton, full-term gestational birth (≥ 37 completed weeks of gestation), with a birth weight of ≥ 2.5 kg and ≤ 4.5 kg
4. Toddler's parent(s)/guardian is of legal age of consent, has sufficient command of English language to complete the informed consent and other study documents, and is willing and able to fulfill the requirements of the study protocol
5. Toddler's parent(s)/guardian can be contacted directly by telephone or email throughout the study

Exclusion Criteria:

Toddlers who exhibit one or more of the following criteria are excluded from enrollment in the study:

1. Chronic infectious, metabolic, genetic illness or other disease including any condition that impacts feeding or may impact outcome measures
2. Known or suspected cows' milk protein intolerance / allergy or severe food allergies that impact diet
3. Toddlers fed vegan, vegetarian, or vegetarian plus fish diets
4. Cognitive or developmental disorders
5. Breast milk used exclusively in place of all other milk, and/or milk alternatives at 17-18 months (GUM & cows' milk group exclusion only, eligible for population group)
6. Consuming supplement(s) of relevance to the study outcome relating diet to status, docosahexaenoic acid (DHA), lutein, and/or choline in amounts >%10 requirements
7. Toddlers or toddlers' family who in the Investigator's judgment cannot be expected to comply with the protocol or study procedures

Ages: 17 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Comparison of blood nutrient markers after 6 months of intervention | 6 months
  To compare blood status of the key nutrients of interest after 180 days of intervention in toddlers randomized in a double-blind manner to Test GUM compared to standard GUM. A non-randomized group for comparison will drink either cows' milk (comparator group) as currently recommended by Health Canada, or participate in a reference group with no drinking or feeding interventions.

SECONDARY OUTCOMES:
Executive function and language development | 6 months
  To assess the effect of milk/drink on measures of neurological development. Standard and validated tools will be used in the assessment including Bayley Scales of Infant Development III
Visual acuity with Teller Acuity Cards | 6 months
  To characterize the effects of milk/drink on visual acuity
Behavioural development | 6 months
  To characterize the effects of milk/drink on behavioural development using standard questionnaires including the Child Behaviour Checklist (CBCL)
Dietary nutrient intake | 6 months
  To characterize effects of milk/drink on dietary intake of energy, macronutrients and key nutrients of interest using the Food Frequency Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Lamers, PhD, Principal Investigator — University of British Columbia; Tim Oberlander, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Children and Women's Health Centre of British Columbia Branch, Vancouver, Canada

IPD SHARING:
Plan to Share IPD: Undecided